CLINICAL TRIAL: NCT00781859
Title: A Randomized, Placebo Controlled, Double-masked, Multicenter Trial of Microplasmin Intravitreal Injection for Non-surgical Treatment of Focal Vitreomacular Adhesion
Brief Title: Trial of Microplasmin Intravitreal Injection for Non-surgical Treatment of Focal Vitreomacular Adhesion. The MIVI-TRUST (TG-MV-006) Trial.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ThromboGenics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TG-MV-006
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Results first posted 2013-01-28 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-04

CONDITIONS: Vitreomacular Adhesion
MeSH Terms: interventions — microplasmin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 125µg Ocriplasmin (Experimental): 125µg intravitreal injection of ocriplasmin
  Interventions: Drug: 125 µg Ocriplasmin
- Placebo (Placebo Comparator): placebo intravitreal injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 125 µg Ocriplasmin — 125µg ocriplasmin intravitreal injection
  Other Names: microplasmin
  Arms: 125µg Ocriplasmin
Drug: Placebo — Placebo intravitreal injection
  Arms: Placebo

SUMMARY:
The objective of this trial is to evaluate the safety and efficacy of intravitreal microplasmin 125µg dose in subjects wiht focal vitreomacular adhesion.

ELIGIBILITY:
Inclusion Criteria:

* Presence of focal vitreomacular adhesion (i.e., central vitreal adhesion within 6mm Optical Coherence Tomography (OCT) field surrounded by elevation of the posterior vitreous cortex) that in the opinion of the Investigator is related to decreased visual function (such as metamorphopsia, decreased visual acuity, or other visual complaint)

Exclusion Criteria:

* Any evidence of proliferative retinopathy (including Proliferative Diabetic Retinopathy (PDR) or other ischemic retinopathies involving vitreoretinal vascular proliferation) or exudative Age-Related Macular Degeneration (AMD) or retinal vein occlusion in the study eye.
* Subjects with any vitreous hemorrhage or any other vitreous opacification which precludes either of the following: visualization of the posterior pole by visual inspection OR adequate assessment of the macula by either OCT and/or fluorescein angiogram in the study eye.
* Subjects with macular hole diameter > 400 μm in the study eye.
* Aphakia in the study eye.
* High myopia (more than 8D) in study eye (unless prior cataract extraction or refractive surgery that makes refraction assessment unreliable for myopia severity approximation, in which case axial length >28 mm is an exclusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2008-12; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - Retinal Consultants of AZ, Phoenix, Arizona
  - Assocaited Retina Consultants, Ltd., Phoenix, Arizona
  - Retina Centers, P.C., Tucson, Arizona
  - Retina Vitreous Associate Medical Group, Beverly Hills, California
  - VMR Institute, Huntington Beach, California
  - Jules Stein Eye Institute/UCLA, Los Angeles, California
  - Southern California Desert Retina Consultants, Palm Springs, California
  - Retinal Consultants Medical Group, Sacramento, California
  - Rocky Mountain Lions Eye Institute, Aurora, Colorado
  - Colorado Retina Associates, PC, Denver, Colorado
  - National Ophthalmologic Research Institute, Fort Meyers, Florida
  - University of Miami-Bascom Palmer Eye Institute- Palm Beach, Palm Beach, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, PC, Augusta, Georgia
  - Rush University Med. Ctr, Chicago, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - Univ. Of Kentuck/Kentucky-Clinic/Dept of Ophthal & VS, Lexington, Kentucky
  - Maine Vitreoretinal Consultants, LLC, PA, Bangor, Maine
  - National Retina Institute, Towson, Maryland
  - University of Michigan-Kellogg Eye Center, Ann Arbor, Michigan
  - Kresge Eye Institute, Detroit, Michigan
  - Vitreo-Retinal Associates, Grand Rapids, Michigan
  - Associated Retina Consultants, Royal Oak, Michigan
  - Vitroretinal Surgery PA, Minneapolis, Minnesota
  - Retina Vitreous Centre, PA, New Brunswick, New Jersey
  - Retina Association of NJ, Teaneck, New Jersey
  - New York Eye and Ear Infirmary, New York, New York
  - Columbia University - Harkness Eye Institute, New York, New York
  - Retina Vitreous Surgeons of Central NY, New York, New York
  - Duke Eye Center, Durham, North Carolina
  - Caroline Eye Associates, Southern Pines, North Carolina
  - Wake Forest University Eye Center, Winston-Salem, North Carolina
  - Retina Association of Cleveland, Lakewood, Ohio
  - Pennsylvania Retina Specialists, P.C., Camp Hill, Pennsylvania
  - Allegheny Ophthalmic & Orbital Associates, PC, Pittsburgh, Pennsylvania
  - Souteastern Retina Associates, Kingsport, Tennessee
  - Austin Retina Associates, Austin, Texas
  - Vitroretinal Consultants, Houston, Texas
  - Valley Retina Institute, P.A., McAllen, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas

REFERENCES:
- [Derived] Varma R, Haller JA, Kaiser PK. Improvement in Patient-Reported Visual Function After Ocriplasmin for Vitreomacular Adhesion: Results of the Microplasmin for Intravitreous Injection-Traction Release Without Surgical Treatment (MIVI-TRUST) Trials. JAMA Ophthalmol. 2015 Sep;133(9):997-1004. doi: 10.1001/jamaophthalmol.2015.1746. PMID 26068086
- [Derived] Folgar FA, Toth CA, DeCroos FC, Girach A, Pakola S, Jaffe GJ. Assessment of retinal morphology with spectral and time domain OCT in the phase III trials of enzymatic vitreolysis. Invest Ophthalmol Vis Sci. 2012 Oct 25;53(11):7395-401. doi: 10.1167/iovs.12-10379. PMID 23033391
- [Derived] Stalmans P, Benz MS, Gandorfer A, Kampik A, Girach A, Pakola S, Haller JA; MIVI-TRUST Study Group. Enzymatic vitreolysis with ocriplasmin for vitreomacular traction and macular holes. N Engl J Med. 2012 Aug 16;367(7):606-15. doi: 10.1056/NEJMoa1110823. PMID 22894573
- [Derived] DeCroos FC, Toth CA, Folgar FA, Pakola S, Stinnett SS, Heydary CS, Burns R, Jaffe GJ. Characterization of vitreoretinal interface disorders using OCT in the interventional phase 3 trials of ocriplasmin. Invest Ophthalmol Vis Sci. 2012 Sep 21;53(10):6504-11. doi: 10.1167/iovs.12-10370. PMID 22879421

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient was recruited on 30 Dec 2008 and last patient completed the study on 17 March 2010
Groups:
- Ocriplasmin 125µg: 125µg ocriplasmin intravitreal injection
- Placebo: Intravitreal injection of placebo
Period: Overall Study
Arm/Group | Ocriplasmin 125µg | Placebo
Started | 219 | 107
Completed | 200 | 98
Not Completed | 19 | 9
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 8 | 4
Not completed — Lost to Follow-up | 6 | 3
Not completed — Death | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ocriplasmin 125µg: 125µg microplasmin intravitreal injection
- Total: Total of all reporting groups
Arm/Group | Ocriplasmin 125µg | Placebo | Total
Number analyzed (Participants) | 219 | 107 | 326
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (10.25) | 71.1 (10.04) | 71.3 (10.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 59 | 207
  Male | 71 | 48 | 119

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Nonsurgical Resolution of Focal Vitreomacular Adhesion at Day 28.
Description: The primary efficacy endpoint was the proportion of subjects with nonsurgical resolution of focal vitreomacular adhesion at Day 28 post-injection, as determined by masked Central Reading Center (CRC) Optical Coherence Tomography (OCT) evaluation. Any subjects who had a creation of an anatomical defect (i.e. retinal hole, retinal detachment) that resulted in loss of vision or that required additional intervention were not counted as successes for this primary endpoint.
Time Frame: Day 28
Population: Intention-To-Treat (ITT), Last Observation Carried forward (LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Ocriplasmin 125µg | Placebo
Number analyzed (Participants) | 219 | 107
percentage of participants | 27.9 | 13.1
Statistical Analysis 1: Comparison: Ocriplasmin 125µg vs Placebo; Test type: Superiority or Other; p = 0.003, Fisher Exact — comparing placebo and ocriplasmin; Odds Ratio (OR) = 2.56, 95% CI 2-sided [1.32 to 5.24]

2. Secondary Outcome: Proportion of Subjects With Total Posterior Vitreous Detachment (PVD) at Day 28
Description: The key secondary endpoint of this study was the proportion of subjects with total Posterior Vitreous Detachment (PVD) at Day 28, as determined by masked Investigator assessment of B-scan ultrasound.
Time Frame: Day 28
Population: Intention-To-Treat (ITT, Last Observation Carried Forward (LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Ocriplasmin 125µg | Placebo
Number analyzed (Participants) | 219 | 107
percentage of participants | 16.4 | 6.5

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs)/Serious Adverse Events (SAEs) were collected from injection day up to 6 months post injection.
Description: AEs/SAEs were assessed by the investigator at all study visits.
Arm/Group | Ocriplasmin 125µg | Placebo
Serious Adverse Events (participants affected / at risk) | 32/220 | 13/106
Other Adverse Events (participants affected / at risk) | 127/220 | 35/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocriplasmin 125µg (N=220) | Placebo (N=106)
Macular hole (Eye disorders) | 16 (17) | 11 (11)
Retinal detachment (Eye disorders) | 2 (2) | 2 (3)
Maculopathy (Eye disorders) | 3 (3) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrahge (Gastrointestinal disorders) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebral hemorrahge (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocriplasmin 125µg (N=220) | Placebo (N=106)
Vitreous floaters (Eye disorders) | 44 (49) | 10 (10)
Conjunctival Hemorrhage (Eye disorders) | 34 (35) | 14 (14)
Photopsia (Eye disorders) | 37 (40) | 4 (4)
Eye pain (Eye disorders) | 34 (39) | 6 (6)
Vision blurred (Eye disorders) | 25 (27) | 5 (7)
Visual impairment (Eye disorders) | 21 (23) | 3 (3)
Visual acuity reduced (Eye disorders) | 14 (15) | 6 (6)
Photophobia (Eye disorders) | 14 (14) | 0 (0)
Retinal edema (Eye disorders) | 13 (14) | 1 (1)
Intraocular pressure incresed (Eye disorders) | 9 (9) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less